CLINICAL TRIAL: NCT00866996
Title: A Multi-center Randomized Parallel Group Study Evaluating Treatment Outcomes of Concerta (Extended Release Methylphenidate) and Strattera (Atomoxetine) in Children With Attention-deficit/Hyperactivity Disorder
Brief Title: Community-based Study Comparing Extended-release Methylphenidate and Atomoxetine in Children With Attention-deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR008329
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention deficit hyperactivity disorder; Methylphenidate; Atomoxetine; Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Methylphenidate extended-release; Atomoxetine

SUMMARY:
The purpose of this study was to better understand the treatment outcomes of extended-release methylphenidate and atomoxetine in children with attention-deficit hyperactivity disorder (ADHD) as evaluated by physicians and parents in a community setting.

DETAILED DESCRIPTION:
Methylphenidate and atomoxetine are available for the treatment of ADHD in children. Methylphenidate is thought to block the reuptake of norepinephrine and dopamine into the presynaptic neuron and increase the release of these monamines into the extraneuronal space. The mechanism by which atomoxetine produces its therapeutic effect is thought to be related to selective inhibition of the presynaptic norephinephrine transporter. This was a multi-center, randomized, open-labeled, parallel design study of extended-release methylphenidate and atomoxetine in children aged 6 to 12 years with ADHD as evaluated by physicians and parents. Children were randomly assigned (2:1, respectively) to 3 weeks of treatment with extended-release methylphenidate or atomoxetine. Physicians evaluated treatment using the ADHD Rating Scale (ADHD-RS) and the Clinical Global Impression-Improvement of Illness scale (CGI-I). Assessments were made prior to beginning treatment (screening), at a telephone interview 1 week after beginning treatment, at a clinic visit 2 weeks after beginning treatment, and at the final clinic visit (3 weeks). Parents assessed treatment using the Parent Satisfaction Questionnaire (PSQ) from treatment days 2 to 13 and at the clinical visit 3 weeks after beginning treatment. The questions of interest included whether there is a difference between treatment in the improvement of behavior and the timing of such differences. Vital signs, height, and weight were also recorded as were adverse events. Study drug was to be taken orally once each day. Patients randomly assigned to extended-release methylphenidate began treatment with 18 mg/day. Patients randomly assigned to atomoxetine began treatment with 0.5 mg/kg/day. The study medication was to be titrated as considered appropriate by the patient's physician. The duration of treatment was 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the DSM-IV criteria for a primary diagnosis of ADHD of any subtype (may have been newly diagnosed with ADHD and not on treatment)
* score of 24 or higher on the ADHD Rating Scale (ADHD-RS) at screening
* physician must have rated the patient as "Moderately ill" or worse on the CGI-S at screening
* children may have been enrolled who were not receiving adequate treatment for ADHD (based on clinical judgment in consultation with the parent)
* children must have been washed-out of their current treatment a minimum of 3 days or 5 half lives of the medication whichever was longer
* and the child and parent must have given written informed consent, and assent, where applicable.

Exclusion Criteria:

* Female child who had experienced menarche
* presence of eating or substance disorder or co-morbid psychiatric condition other than oppositional defiant disorder
* history of seizure, tic disorder, mental retardation, severe developmental disorder (i.e. severe cerebral palsy, autism) or family history of Tourette's Disorder
* required medications as excluded by the package inserts for Concerta or Strattera
* diagnosed with hyperthyroidism or glaucoma
* and known non-responders to treatments indicated for ADHD.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1323 (Actual)
Dates: Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Observed and change from baseline measures for ADHD-RS total scores will be summarized by descriptive statistics and analyzed by repeated measures of analysis of covariance.

SECONDARY OUTCOMES:
CGI-I and each PSQ item separately were summarized by descriptive statistics and frequency distributions. Treatment effects were tested by chi-square statistics. Onset of effect was assessed by PSQ on Days 2 to 13.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Result] Kemner JE, Starr HL, Ciccone PE, Hooper-Wood CG, Crockett RS. Outcomes of OROS methylphenidate compared with atomoxetine in children with ADHD: a multicenter, randomized prospective study. Adv Ther. 2005 Sep-Oct;22(5):498-512. doi: 10.1007/BF02849870. PMID 16418159
- [Result] Starr HL, Kemner J. Multicenter, randomized, open-label study of OROS methylphenidate versus atomoxetine: treatment outcomes in African-American children with ADHD. J Natl Med Assoc. 2005 Oct;97(10 Suppl):11S-16S. PMID 16350601
- See also: Community-based study comparing extended-release methylphenidate and atomoxetine in children with attention-deficit hyperactivity disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1090&filename=CR008329_CSR.pdf